CLINICAL TRIAL: NCT06245161
Title: Efficacy of Computer Controlled Intraosseous Anesthesia in Pediatric Dental Patients (Randomized Controlled Clinical Trial)
Brief Title: Efficacy of Computer Controlled Intraosseous Anesthesia in Pediatric Dental Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0588-01/2023
Record Dates: First submitted 2023-10-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2023-10

CONDITIONS: Irreversible Pulpitis; Tooth Extraction
Keywords: Intraosseous anesthesia; Computer-controlled injection; pain management; dental anesthesia; pediatric dentistry
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: 120 children eligible for the study will be divided into: Group I (restorative group): includes 60 quadrants, each have at least one primary molar indicated for restorative treatment or vital pulp therapy. It will be subdivided into 4 subgroups, each consists of 15 quadrant (upper and lower) allocated to Intra-osseous Anesthesia by QuickSleeper5 for the test groups or to infiltration or IANB in the control group
  Group II (extraction group): includes 60 primary molars indicated for extraction. It will be subdivided into 4 subgroups; according either maxillary or mandibular primary molar is indicated for extraction, using Intra-osseous Anesthesia by QuickSleeper5 for the test groups ,or infiltration or IANB in the control group
Who Masked: Participant
Masking Description: participants are blinded to the group assignment, as their visual field is blocked during needle adminstration in both groups, and the Audible sounds of the QuickSleeper5 will be mimicked in the control group.
  The operator will not be blinded to the type of the anesthesia administered due to different devices to be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- • Group IA (Experimental): 15 maxillary quadrants each have at least one primary molar indicated for restorative treatment or vital pulp therapy, allocated to Intra-osseous Anesthesia by QuickSleeper5.
  Interventions: Device: Quicksleeper5
- • Group IB (Active Comparator): 15 maxillary quadrants each have at least one primary molar indicated for restorative treatment or vital pulp therapy, allocated to infiltration anesthesia
  Interventions: Device: conventional anesthesia
- • Group IC (Experimental): 15 Mandibular quadrants each have at least one primary molar indicated for restorative treatment or vital pulp therapy, allocated to Intra-osseous Anesthesia by QuickSleeper5.
  Interventions: Device: Quicksleeper5
- • Group ID (Active Comparator): 15 mandibular quadrants each have at least one primary molar indicated for restorative treatment or vital pulp therapy, allocated to inferior alveolar nerve block (IANB) anesthesia
  Interventions: Device: conventional anesthesia
- • Group IIA (Experimental): 15 maxillary primary molars indicated for extraction allocated to Intra-osseous Anesthesia by QuickSleeper5
  Interventions: Device: Quicksleeper5
- • Group IIB (Active Comparator): 15 maxillary primary molars indicated for extraction allocated to Infiltration anesthesia
  Interventions: Device: conventional anesthesia
- • Group IIC (Experimental): 15 Mandibular primary molars indicated for extraction, allocated to Intra-osseous Anesthesia by QuickSleeper5
  Interventions: Device: Quicksleeper5
- • Group IID (Active Comparator): 15 Mandibular primary molars indicated for extraction, allocated to inferior alveolar nerve block (IANB) anesthesia.
  Interventions: Device: conventional anesthesia

INTERVENTIONS:
Device: Quicksleeper5 — intraosseous anesthesia for dental treatment
  Arms: • Group IA; • Group IC; • Group IIA; • Group IIC
Device: conventional anesthesia — inferior alveolar nerve block for treating mandibular molars infiltration anesthesia for treating maxillary molars
  Arms: • Group IB; • Group ID; • Group IIB; • Group IID

SUMMARY:
To evaluate the effectiveness of intra-osseous anesthesia using Quicksleepr5 in pain elimination during dental treatment in maxillary and mandibular primary molars, compared to conventional anesthesia.

DETAILED DESCRIPTION:
The study will be an eight-armed randomized controlled trial, parallel design. A total of 120 pediatric dental patients aged from 5 to 9 years with good health, will be selected from the Pediatric Dentistry and Dental Public Health Department clinic, Faculty of Dentistry, Alexandria University, Egypt. They will be recruited among those who need local anesthesia to perform either quadrant restorative treatment or extraction of their primary molars. Participants will be allocated into 2 groups according to the local anesthetic technique to be used. Children in the test group will receive intraosseous anesthesia using QuickSleeper5, while inferior alveolar nerve block or infiltration anesthesia will be used for those who are in the control group. All the procedures will be videotaped. Pain response upon needle prick and dental treatment will be assessed subjectively using the visual analogue scale, and objectively using Face, Leg, Activity, cry, Consolability scale. Physiological parameters will also be recorded to determine pain reaction. Efficacy, latency period and duration of anesthesia will be recorded for both injection techniques. Child behaviour toward dental treatment in both injection techniques will be evaluated using Frankl rating scale. Dental anxiety of pediatric patients will be evaluated from the videotapes using VENHAM Clinical Anxiety Scale. Postoperative assessment for the occurrence of any adverse events is planned.

ELIGIBILITY:
Inclusion Criteria:

* Cooperative children during preoperative assessments.
* Patients selected in the restorative group: presenting with at least one primary molar indicated for restorative treatment or vital pulp therapy, after thorough clinical and radiographic examination.
* Patients selected in the extraction group: presenting with at least one primary molar indicated for extraction.

Exclusion Criteria:

* Any physical or mental disability, or psychological problems.
* Immunocompromised patients.
* Hypersensitivity to local anesthetic drugs used
* History of previous dental local anesthesia.
* Taking analgesics or other medications that would alter the child behavior or awareness of pain 12- hours pre-operative

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of Pain Reaction objectively | 1- Preoperatively phase (baseline) 2- During LA administration. 3-During dental treatment: Rubber dam placement and tooth preparation Or tooth extraction
  Pain response will be assessed using Face, Legs, Activity, Cry Consolability (FLACC) scale
Assessment of Pain Reaction subjectively | 1-Post injection phase (1- minute). 2- Post treatment phase (10 minutes)
  it will done by the child using Face version of Visual Analogue Scale.
Child dental anxiety | 1-Preoperative phase (baseline) 2- During local anesthesia administration 3-During dental treatment (restorative or extraction)
  It will be assessed using VENHAM Clinical Anxiety Scale

SECONDARY OUTCOMES:
Local anesthesia effect | 30 minutes postoperatively
  efficacy of anesthesia (using efficacy scale by Sixou et al )
Assessment of occurrence of adverse events | follow up 24 hour postoperatively
  the occurrence of self-inflicted injury, pain at injection site or trismus, or any adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: sara quritum, Principal Investigator — Alexandria Univeristy
Locations (1):
- Alexandria University- Faculty of Dentistry, Alexandria, Alexandroa, Egypt